CLINICAL TRIAL: NCT05088369
Title: A First-in-human, Double-blind, Placebo-controlled, Phase 1 Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Intravenous Doses of HM201 (Pegylated Human Adrenomedullin) in Healthy Subjects (Adults)
Brief Title: Assessment of the Safety, Tolerability, and Pharmacokinetic of HM201
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syneos Health (Other)
Collaborators: Himuka AM Pharma Corp. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM201-AUS-001
Record Dates: First submitted 2021-10-12; First posted 2021-10-21 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Ulcerative Colitis; Crohn's Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Intervention Model Description: SAD & MAD study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be conducted as a double-blind study. All subjects and clinical personnel will involved in the collection, monitoring, revision, safety and adverse events will be blinded in regards to the subject's treatment assigned of HM201 or the HM201 placebo. All personnel affecting the outcome of the study's treatment assignment will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SAD Cohorts 1 to 4: Participants receiving HM201 (Experimental): Each SAD cohort participant will be randomized to receive 1 of 4 escalating doses (0.01 mg/kg (2 nmol/kg); 0.03 mg/kg (5 nmol/kg); 0.06 mg/kg (10 nmol/kg); 0.12 mg/kg (20 nmol/kg).
  Interventions: Drug: HM201
- SAD Cohorts 1 to 4: Participants Receiving Placebo (Placebo Comparator): Each SAD cohort participant will be randomized to receive placebo.
  Interventions: Drug: Placebo
- MAD Cohorts 1 to 4: Participants Receiving HM201 (Experimental): Each MAD cohort participant will be randomized to receive a once a week dose of 1 of 4 escalating doses (0.01 mg/kg (2 nmol/kg); 0.03 mg/kg (5 nmol/kg); 0.06 mg/kg (10 nmol/kg), 0.12 mg/kg (20 nmol/kg) for 4 weeks.
  Interventions: Drug: HM201
- MAD Cohorts 1 to 4: Participants Receiving Placebo (Placebo Comparator): Each MAD cohort participant will be randomized to receive placebo once a week for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HM201 — HM201 will be administered intravenously.
  Other Names: Pegylated human adrenomedullin
  Arms: SAD Cohorts 1 to 4: Participants receiving HM201
Drug: Placebo — Placebo will be administered intravenously.
  Other Names: Matching Placebo
  Arms: SAD Cohorts 1 to 4: Participants Receiving Placebo
Drug: HM201 — HM201 will be administered intravenously.
  Other Names: Pegylated human adrenomedullin
  Arms: MAD Cohorts 1 to 4: Participants Receiving HM201
Drug: Placebo — Placebo will be administered intravenously.
  Other Names: Matching Placebo
  Arms: MAD Cohorts 1 to 4: Participants Receiving Placebo

SUMMARY:
This will be a single centre, Phase 1, Placebo-controlled, Randomized, Doubleblind, SAD & MAD Study to Assess the Safety, Tolerability and PK of HM201 in Healthy Subjects.

DETAILED DESCRIPTION:
Objective of the study is to assess the safety, tolerability, and PK of single and multiple intravenous administration of HM201. The study design consists of a SAD study of 4 cohorts, 8 subjects each cohort and a different dose level per cohort. In each cohort 2 will receive the placebo while rest of group will be administered with HM201. A total of 32 subjects are planned for the SAD study.

MAD part will begin after cohort 1 and 2 of SAD is completed. MAD will consist of 8 subjects; 2 will receive the placebo while 6 will be administered with HM201. MAD will be conducted in a dose escalation manner with 4 weekly doses administered to all subjects. One randomization scheme will be produced for each cohort separately.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy male or non-childbearing potential female
2. BMI ≥18.0 and ≤32.0 kg/m2
3. Good health based on past medical history, medication use, vital signs and physical exam.
4. Normal renal and hepatic function.
5. Female partners of child bearing potential must agree to use contraception.

Key Exclusion Criteria:

1. Clinically significant medical history.
2. Significant drug allergy.
3. Use of experimental drug within 3 months prior.
4. Previously received HM201, AM and other derivatives.
5. History of old myocardial infarction.
6. Diagnosed with malignant tumor or history of treatment for malignant tumor.
7. History of drug or alcohol abuse.
8. Use of omitted medicines or substance opposing objective of study.
9. COVID19 vaccine administered within 14 days of initiation of investigational product or if to receive additional dose within 30 days of investigational product administration.
10. Use of tobacco/nicotine in excess of ≥ 5 cigarettes a day and unable or unwilling to prohibit smoking during admission to site.
11. Daily consumption of more than 1L of caffeine/xanthine beverage which cannot be discontinued more than 24 hours prior to dosing of investigational product and/or ECG measurement.
12. Regular use of nutraceuticals (e.g., St. John's wort, ginseng, ginkgo biloba, Chinese herbs, and melatonin) within 1 week before administration of investigational product.
13. Donation of plasma or platelet or 200 mL of whole blood within 4 weeks or 400 mL whole blood within 3 months before administration of investigational product.
14. Clinically relevant findings in ECG.
15. Systolic blood pressure below 100 mmHg or above 140 mmHg at screening.
16. Diastolic blood pressure above 90 mmHg at screening.
17. Heart rate below 40 beats/min or above 100 beats/min at screening.
18. Symptom of orthostatic hypotension is found at screening or before investigational product administration (Day -1).
19. Hepatitis B virus surface antigen (HBsAg), hepatitis B virus core antibody (HBcAb) hepatitis C virus antibodies (anti-HCV) or human immunodeficiency virus (HIV) antigen and antibody at screening.
20. Positive to syphilis.
21. Positive to urine drug test.
22. Positive alcohol breath test.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Number and percentage of treatment-emergent adverse event, serious adverse event and discontinuation. | Up to 15 days post last infusion for both SAD & MAD

SECONDARY OUTCOMES:
Plasma concentrations of HM201 | SAD: Up to Day 15. MAD: Up to Day 36
Pharmacokinetic assessment 1 | SAD: Up to Day 15. MAD: Up to Day 36
  Area under the plasma concentration versus time curve (AUC)
Pharmacokinetic assessment 2 | SAD: Up to Day 15. MAD: Up to Day 36
  Peak Plasma Concentration (Cmax)
Pharmacokinetic assessment 3 | SAD: Up to Day 15. MAD: Up to Day 36
  Time of peak plasma concentration (Tmax)
Pharmacokinetic assessment 4 | MAD: Up to Day 36
  Concentration at the last planned timepoint prior to dosing (Ctrough)
Pharmacokinetic assessment 5 | SAD: Up to Day 15. MAD: Up to Day 36
  Mean residence time (MRT)
Pharmacokinetic assessment 6 | SAD: Up to Day 15. MAD: Up to Day 36
  Drug clearance (CL) & Clearance at steady state (CLss)
Pharmacokinetic assessment 7 | SAD: Up to Day 15. MAD: Up to Day 36
  Volume of distribution at steady state (Vss) & during terminal phase (VZ)
Pharmacokinetic assessment 8 | SAD: Up to Day 15. MAD: Up to Day 36
  Half life (T1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Kristi McLendon, MD, Principal Investigator — Nucleus Network Pty Ltd.
Locations (1):
- Nucleus Network Pty Ltd, Herston, Queensland, Australia